CLINICAL TRIAL: NCT02805010
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Pharmacokinetics, Safety and Tolerability of Single Dose of Abatacept 125mg Administered Subcutaneously in Chinese Healthy Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability Study of Single Dose of Abatacept 125mg Administered Subcutaneously
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-126-I
Record Dates: First submitted 2016-06-12; First posted 2016-06-17 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous(SC) Abatacept (Experimental)
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Abatacept — On Day 1, subjects will receive a single SC dose of abatacept 125mg
  Other Names: Orencia
  Arms: Subcutaneous(SC) Abatacept
Other: Placebo — On Day 1, subjects will receive a single SC dose of placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to assess the single dose PK, safety, tolerability and immunogenicity of abatacept 125mg administered SC in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are willing to participate in this study and signed informed consent;
* Healthy subjects, as determined by no clinically significant deviation from normal in medical history, physical examination, Electrocardiograph（ECG）, and clinical laboratory determinations;
* Body weight for male must be≥50 kg, for female be≥45 kg, and all subjects must be ≤100kg;
* Body mass index (BMI) is 19-26 kg/m2 (boundary value included), [BMI = body weight (kg) / height (m)2];
* Men and women, 18-45 years old (boundary value included);
* Women of child bearing potential (WOCBP) must be using the adequate method of contraception to avoid pregnancy throughout the study, for 4 weeks before and for up to 10 weeks after administration of abatacept, male subjects of childbearing potential must be using an adequate method of contraception throughout the study and for up to 10 weeks after administration of investigational product in such a manner that risk of pregnancy is minimized;

  * WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal. Post-menopausal is defined as: Amenorrhea ≥ 12 consecutive months without another cause, or for women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL;
  * Women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential;
* WOCBP must have a negative serum pregnancy test within 24 hours prior to study medication administration.

Exclusion Criteria:

* WOCBP and males subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for up to 10 weeks after administration of the study medication;
* Women who are pregnant or breast-feeding;
* History or concurrent diseases of central nervous system, cardiovascular system, renal, hepatic, digestive tract, respiratory system, metabolism and musculoskeletal system. (including but not limited to arrhythmia, bradycardia, hypotension, coronary heart disease, bronchial asthma, diabetes, hyperthyroidism, Parkinson's disease, epilepsy, shaking palsy, cancer, etc.). Or any other diseases or physiological abnormalities, which might affect study results;
* Any major surgery within 4 weeks of enrollment;
* Splenectomized subjects;
* Exposed to any investigational medication within 3 months of enrollment, or plan to receive other investigational medication during the study;
* Donation of blood or plasma within 3 months of enrollment, or plan to donate blood or plasma during the study or within one month after the end of the study;
* Blood transfusion within 4 weeks prior to enrollment;
* Subjects who is a current smoker (defined as individuals who smoked for more than 6 months, and smoked for ≥ 5 cigarettes per day before screening), ≥ 3 cups of coffee or other coffee drinks or ≥ 5 cups of tea per day;
* Subjects who have a history of drug or alcohol abuse;
* Subjects with tuberculosis (TB) risk, specially:

  * Having clinical, imaging or lab test evidences of current active or latent pulmonary tuberculosis;
  * Having active pulmonary tuberculosis during the past 3 years, even if had been treated;
  * Having history of active pulmonary tuberculosis more than 3 years ago, unless the appropriate duration and types of anti-tuberculosis drug is well documented.
* Subjects with herpes zoster that resolved less than 2 months prior to enrollment;
* Subjects who had any acute or chronic bacterial infection in the previous 3 months prior to enrollment;
* Subjects who have acute and latent bacterial and viral infection (as assessed by the investigator) at the time of enrollment, including subjects with evidence of Human Immunodeficiency Virus (HIV) infection;
* Subjects who have mental or physical disability;
* Subjects who have any surgical and medical conditions, which might be harmful if subjects participate in the study, or which might change the absorption, distribution, metabolism and excretion of investigational medication;
* Heart beat rate <50 beats /min or >100 beats /min (heart rates should be measured after a brief period of rest, at least 5 minutes.), systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg, body temperature (forehead)>37.6℃;
* Hgb < LLN (lower limit of normal), the absolute neutrophil count (ANC) <1.5×10^9/L, platelets <100×10^9/L; bilirubin > ULN (upper limit of normal), serum creatinine > ULN ; glutamic oxaloacetic transaminase (AST) > ULN, glutamic pyruvic transaminase (ALT) > ULN;
* Subject who have active infection, or positive for hepatitis-B surface antigen (HBs-Ag), hepatitis-C antibody (HCV-Ab), or HIV-Ab;
* Positive urinalysis for protein, or other abnormal urinalysis tests which were judged to have clinical significance by investigators;
* History of drug allergy, postural hypotension, or idiopathic allergy;
* Prior exposure to abatacept (CTLA4-Ig), belatacept (LEA29Y) or any leukocyte depleting agent;
* Use of any prescription drugs within 4 weeks (or 5 half-lives, whichever is longer) prior to enrollment, Use of any OTC medications and herbal preparations within 1 week prior to enrollment, unless the medical monitoring shows that the drug has been cleared;
* Vaccination with any live vaccine within 4 weeks prior to study medication administration on Day 1;
* Administration of oral polio vaccine to subject or house hold contacts during the course of study;
* Prisoners or subjects who are involuntarily incarcerated;
* Subjects who are compulsorily detained for treatment either a psychiatric or physical (e.g., infectious disease) illness.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Day1 to Day71
Area Under the Curve (AUC) | Day1 to Day71
Half-life period (T1/2) | Day1 to Day71
Time to peak (Tmax) | Day1 to Day71

SECONDARY OUTCOMES:
Adverse event (AE) | Signed Informed consent form (ICF) to Day 71
anti-abatacept antibodies | Day1 to Day 71
Anti cytotoxic T lymphocyte-associated antigen-4(CTLA-4) antibodies | Day1 to Day 71

IPD SHARING:
Plan to Share IPD: No